CLINICAL TRIAL: NCT00594997
Title: A School-Based Intervention to Reduce Lyme Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Nancy Shadick, Associate Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2004P001033
Record Dates: First submitted 2008-01-07; First posted 2008-01-16 (Estimated); Results first posted 2021-04-06 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Lyme Disease
Keywords: Lyme disease; educational intervention for children; tick borne illness; prophylactic therapy in children; Self-efficacy; tick prevention; tick avoidance; health behavior modification
MeSH Terms: conditions — Lyme Disease | interventions — Educational Status; Lead

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Education (Experimental): Students who receive an educational intervention which consists of a 45 minute interactive presentation as well as a 30 minute health education entertainment by a juggler.
  Interventions: Behavioral: Education
- Control (Active Comparator): Students who fill out pre and post surveys and receive the intervention after the post-survey
  Interventions: Behavioral: Control (pre and post surveys)

INTERVENTIONS:
Behavioral: Education — Students receive an educational intervention delivered by a member of our staff in conjunction with the teacher as well as a health education entertainer
  Arms: Education
Behavioral: Control (pre and post surveys) — Students fill out a pre and post survey and then receive the same intervention given to the controls.
  Arms: Control

SUMMARY:
Our overall purpose of this study is evaluate whether a short in-class Lyme Disease education program based on social learning theory and the Health Belief Model can impact a child's knowledge, attitude, and preventive behavior.

1. Deliver an educational program in schools to promote personal protective practices, encourage early disease detection and modify residential habitats to reduce tick density.

3. Evaluate the program's efficacy by comparing the acceptability and practice of precautionary behavior, tick density in residential areas and rates of Lyme disease between groups using primary and surveillance data sources Evaluate the contribution of knowledge, attitudes, and parental involvement to children's adoption of prevention strategies.

Hypothesis

The community intervention will reduce the incidence of Lyme disease among children and families living in endemic areas by increasing the practice of precautionary behavior and reducing tick density in residential areas. Specifically, we hypothesize that:

1. The educational intervention will reduce the incidence of Lyme disease among children and families living in an endemic area.
2. The educational intervention will improve the childrens' self-confidence (behavioral self-efficacy), intention to perform, and actual practice of Lyme disease prevention behaviors.

DETAILED DESCRIPTION:
The description of Lyme disease in 1976 and subsequent characterization of its mode of transmission, causative organism and treatment is one of the most remarkable advances in medicine in the last 25 years1-3. Nevertheless, Lyme disease continues to grow as a public health problem4. While Lyme disease affects all age groups, children have one of the highest rates4. Prevention remains a challenge in this group. The Lyme vaccine has been withdrawn from the market in February 20025, 6, and educational strategies among at-risk school children have been inadequately evaluated and none have been institutionalized.

We will target school-aged children living in Nantucket, Dukes County and Essex County. We have collaborated with the teachers and administration in many of the schools. We have collaborated with the teachers and administration in many of the schools.

The intervention will be delivered by a member of our staff in conjunction with the teacher as well as a health education entertainer ('Screaming with Pleasure Productions'). Research assistants will distribute the enrollment questionnaires and "goody" bags. The basic content of the educational message has been designed by Drs. Shadick, Liang, DeJong and the late Dr. Daltroy, and has been used extensively on the Nantucket ferry study and in the "Feel Find Free" Program. The timing takes advantage of the classroom audience, is humorous and entertaining and the message is relevant to anticipated outdoor activities.

Primary Outcome: The educational intervention will reduce the incidence of Lyme Disease among children and families living in an endemic area.

Secondary Outcomes: The educational intervention will improve the children's self-confidence (behavioral self-efficacy), intention to perform, and actual practice of Lyme disease prevention behaviors.

ELIGIBILITY:
Inclusion:

* Child age 7-12 and their parents living in the selected endemic areas

Exclusion:

* No exclusions

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3570 (Actual)
Dates: Start 2004-04; Primary Completion 2006-03 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy A Shadick, MD, MPH, Principal Investigator — Brigham and Women's Hospital

REFERENCES:
- [Background] Daltroy LH, Phillips C, Lew R, Wright E, Shadick NA, Liang MH. A controlled trial of a novel primary prevention program for Lyme disease and other tick-borne illnesses. Health Educ Behav. 2007 Jun;34(3):531-42. doi: 10.1177/1090198106294646. Epub 2007 Apr 27. PMID 17468463
- [Background] Corapi KM, White MI, Phillips CB, Daltroy LH, Shadick NA, Liang MH. Strategies for primary and secondary prevention of Lyme disease. Nat Clin Pract Rheumatol. 2007 Jan;3(1):20-5. doi: 10.1038/ncprheum0374. PMID 17203005
- [Background] Phillips CB, Liang MH, Sangha O, Wright EA, Fossel AH, Lew RA, Fossel KK, Shadick NA. Lyme disease and preventive behaviors in residents of Nantucket Island, Massachusetts. Am J Prev Med. 2001 Apr;20(3):219-24. doi: 10.1016/s0749-3797(00)00315-9. PMID 11275450
- [Background] Shadick NA, Lew RA, Liang MH. Outcomes of Lyme Disease. Ann Intern Med. 2000 Nov 7;133(9):746-747. doi: 10.7326/0003-4819-133-9-200011070-00023. No abstract available. PMID 11074914
- [Background] Shadick NA, Daltroy LH, Phillips CB, Liang US, Liang MH. Determinants of tick-avoidance behaviors in an endemic area for Lyme disease. Am J Prev Med. 1997 Jul-Aug;13(4):265-70. PMID 9236962
- [Derived] Shadick NA, Zibit MJ, Nardone E, DeMaria A Jr, Iannaccone CK, Cui J. A School-Based Intervention to Increase Lyme Disease Preventive Measures Among Elementary School-Aged Children. Vector Borne Zoonotic Dis. 2016 Aug;16(8):507-15. doi: 10.1089/vbz.2016.1942. Epub 2016 Jun 1. PMID 27248436

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Education | Control
Started | 1562 | 2008
Completed | 1562 | 2008
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Education | Control | Total
Number analyzed (Participants) | 1562 | 2008 | 3570
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.1 (1.2) | 9.1 (1.2) | 9.1 (1.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 822 | 1003 | 1825
  Male | 740 | 1005 | 1745
Grade [Number; unit: participants]
  Second Grade | 335 | 489 | 824
  Third Grade | 410 | 514 | 924
  Fourth Grade | 422 | 474 | 896
  Fifth Grade | 393 | 528 | 921
  Missing | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: The Incidence of Lyme Disease Among Children and Families Living in an Endemic Area Using an Educational Intervention
Description: Parents of children were asked at baseline to report any new case of Lyme Disease within the past 12 months. This question was asked again a year later after receiving the educational intervention was given. We then will compare the number of reported Lyme Disease cases at baseline to the number of Lyme disease cases reported a year later. New cases of Lyme Disease had to be confirmed by medical record review.
Time Frame: baseline - 1 year
Population: Number of Lyme cases reported in the intervention and control groups
Measure: Number; unit: Number of cases incident Lyme disease
Groups:
- Education: Number of reported incident cases of Lyme by parents of children who received a 45 minute educational intervention by a health educator.
- Control: The number of incident cases of Lyme reported by parents of students in the control group. These students did not receive the educational intervention.
Arm/Group | Education | Control
Number analyzed (Participants) | 10 | 4
Number of cases incident Lyme disease | 1 | 1

2. Secondary Outcome: The Educational Intervention Will Improve the Children's Self-confidence (Behavioral Self-efficacy), Intention to Perform, and Actual Practice of Lyme Disease Prevention Behaviors.
Description: Three outcome measures, knowledge of LD transmission, self reported tick bite precautionary behaviors and attitudes towards taking precautions were measured. A Lyme Disease knowledge score was created from totaling the number of correct answers on the 6 knowledge questions, ranging from 0-6. A score with a higher value indicated an increase in the desired behavior. These questions were asked before and after the intervention to compared the change from preintervention with postintervention between intervention and control students, adjusted for age, sex and pre-knowledge score. Precautionary behavior outcomes were graded on a linear scale quantifying the amount of practice.
Time Frame: baseline -1 year
Population: Composite knowledge score for intervention and control students post-intervention. Comparing the change in score between intervention and controls between pre and post evaluation.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Education | Control
Number analyzed (Participants) | 1562 | 2008
units on a scale | 1.38 (1.31) | 0.36 (1.30)
Statistical Analysis 1: Comparison: Education vs Control; Test type: Superiority or Other; p < 0.0001, Regression, Linear — p<0.05 threshold for statistical significance

ADVERSE EVENTS:
Description: No adverse events were reported or observed for both the education and control groups
Arm/Group | Education | Control
All-Cause Mortality (participants affected / at risk) | 0/1562 | 0/2008
Serious Adverse Events (participants affected / at risk) | 0/1562 | 0/2008
Other Adverse Events (participants affected / at risk) | 0/1562 | 0/2008

LIMITATIONS AND CAVEATS:
Because all school districts were located in endemic areas for Lyme Disease, there was already a high level of awareness of Lyme Disease.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No